CLINICAL TRIAL: NCT01635153
Title: Randomized Controlled Trial of a Protein-calorie Supplement for HIV-infected Women With Tuberculosis
Brief Title: Effects of a Protein Calorie Supplement in HIV-infected Women With Tuberculosis
Acronym: DarDar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, C. Fordham von Reyn, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DarDar 2-C CPHS 21592 D12221; RO1 503498 (Other: NIH)
Record Dates: First submitted 2012-05-23; First posted 2012-07-09 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: HIV; Tuberculosis
Keywords: HIV; Tuberculosis; Nutrition
MeSH Terms: conditions — Tuberculosis | interventions — Micronutrients

STUDY DESIGN:
Intervention Model Description: Protein-calorie supplement plus micronutrient vs micronutrient alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein calorie supplement plus micronutrient (Active Comparator)
  Interventions: Dietary Supplement: Protein calorie supplement
- Micronutrient alone (Placebo Comparator)
  Interventions: Dietary Supplement: Micronutrient

INTERVENTIONS:
Dietary Supplement: Protein calorie supplement — Fortified porridge with 1062 kcal and 40 gm protein
  Other Names: Dar-uji
  Arms: Protein calorie supplement plus micronutrient
Dietary Supplement: Micronutrient — Dar-vite Multivitamin
  Arms: Micronutrient alone

SUMMARY:
The objective of this randomized, controlled trial is to determine if adding a protein-calorie supplement (PCS) to the standard treatments for tuberculosis (TB) and HIV will improve health outcomes. The investigators will enroll 180 HIV-positive women with newly diagnosed active TB and without prior anti-retroviral therapy (ART). At baseline, the investigators will conduct dietary interviews, measure body composition, randomize subjects to receive a PCS (plus micronutritional supplements [MNS]) or control (MNS only) for the 6-month duration of anti-TB therapy (ATT) plus an additional 2 mos (8 mos total). Subjects will be followed monthly and have CD4 counts at baseline, 2, 8 and 12 months. At 2 months (i.e., at the end of the 4 drug intensive phase of TB treatment and start of the 2 drug continuation phase), all subjects will be started on anti-retroviral therapy (ART) based on Tanzanian Ministry of Health guidelines (currently: AZT/3TC/efavirenz). The primary endpoint will be change in CD4 count after 8 months (i.e., at end of PCS/MNS intervention and 2 months after completion of ATT).

DETAILED DESCRIPTION:
The objective of this randomized, controlled trial is to determine if adding a protein-calorie supplement (PCS) to the standard treatments for tuberculosis (TB) and HIV will improve health outcomes. The investigators will enroll 180 HIV-positive women with newly diagnosed active TB and without prior anti-retroviral therapy (ART). At baseline, the investigators will conduct dietary interviews, measure body composition, randomize subjects to receive a PCS (plus micronutritional supplements [MNS]) or control (MNS only) for the 6-month duration of anti-TB therapy (ATT) plus an additional 2 mos (8 mos total). Subjects will be followed monthly and have CD4 counts at baseline, 2, 8 and 12 months. At 2 months (i.e., at the end of the 4 drug intensive phase of TB treatment and start of the 2 drug continuation phase), all subjects will be started on anti-retroviral therapy (ART) based on Tanzanian Ministry of Health guidelines (currently: AZT/3TC/efavirenz). The primary endpoint will be change in CD4 count after 8 months (i.e., at end of PCS/MNS intervention and 2 months after completion of ATT).

ELIGIBILITY:
Inclusion Criteria:

* female,
* HIV,
* age > 18,
* CD4 > 50,
* BMI>16
* new TB diagnosis,
* not on anti-retroviral therapy,
* residence in Dar es Salaam

Exclusion Criteria:

* current anti-retroviral therapy,
* serious co-morbidities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. von Reyn, MD, Principal Investigator — Dartmouth College; Nyasule Majura-Neke, MD, Study Director — Muhimbili University of Health and Allied Sciences
Locations (1):
- Infectious Disease Centre, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magohe A, Kimario J, Lukmanji Z, Hendricks K, Koethe JR, Neke NM, Tvaroha S, Connor R, Mackenzie T, Waddell R, Maro I, Matee M, Pallangyo K, Bakari M, Horsburgh CR, von Reyn CF. Randomized, controlled trial of a protein-calorie supplement for women coinfected with HIV-TB. Int J Tuberc Lung Dis. 2022 Aug 1;26(8):798-800. doi: 10.5588/ijtld.21.0669. No abstract available. PMID 35898141

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protein Calorie Supplement Plus Micronutrient | Micronutrient Alone
Started | 72 | 79
Completed | 32 | 36
Not Completed | 40 | 43
Not completed — Lost to Follow-up | 40 | 43

BASELINE CHARACTERISTICS:
Population: Non-malnourished women with newly diagnosed TB and newly diagnosed HIV, not on ART at time of enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Protein Calorie Supplement Plus Micronutrient | Micronutrient Alone | Total
Number analyzed (Participants) | 72 | 79 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 79 | 151
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.5 [33.5 to 44.5] | 36 [31 to 43] | 37 [32 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 79 | 151
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 72 | 79 | 151

OUTCOME MEASURES:

1. Primary Outcome: Change in CD4 Count
Description: We will calculate change in CD4 count from start of ART until 6 mos on ART (which is started 2 mos after study enrollment, hence 8 mos after enrollment)
Time Frame: Baseline to 8 months
Population: Women with newly diagnosed TB and newly diagnosed HIV, not on ART
Measure: Mean (Standard Deviation); unit: increase in CD4 cells/mm^3
Arm/Group | Protein Calorie Supplement Plus Micronutrient | Micronutrient Alone
Number analyzed (Participants) | 72 | 79
increase in CD4 cells/mm^3 | 215 (28) | 174 (21)

2. Secondary Outcome: BMI at 6 Months
Description: BMI will be compared between the two treatment groups
Time Frame: baseline to 6 months
Population: Women with newly diagnosed TB and newly diagnosed HIV not on ART
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Protein Calorie Supplement Plus Micronutrient | Micronutrient Alone
Number analyzed (Participants) | 72 | 79
kg/m^2 | 25.4 (5.73) | 24.7 (4.99)

3. Secondary Outcome: Number of Subjects Who Achieve 100 Cell Increase in CD4
Description: Number of subjects in 2 treatment groups who achieve 100 cell increase in CD4 will be compared
Time Frame: baseline to 8 months
Population: Women with newly diagnosed TB and newly diagnosed HIV not yet on ART
Measure: Number; unit: N of subjects with CD4 increase of ≥100
Arm/Group | Protein Calorie Supplement Plus Micronutrient | Micronutrient Alone
Number analyzed (Participants) | 72 | 79
N of subjects with CD4 increase of ≥100 | 25 | 26

ADVERSE EVENTS:
Time Frame: 8 months
Description: Standard definitions
Arm/Group | Protein Calorie Supplement Plus Micronutrient | Micronutrient Alone
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/79
Other Adverse Events (participants affected / at risk) | 0/72 | 0/79

LIMITATIONS AND CAVEATS:
Many patients were lost to follow-up which may interfere with the evaluation of treatment effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No